CLINICAL TRIAL: NCT01331382
Title: Effects of Resveratrol Alone or in Combination With Piperine on Cerebral Blood Flow Parameters and Cognitive Performance in Humans
Brief Title: Cerebral Blood Flow Effects of Resveratrol and Piperine in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Emma Wightman, Northumbria university
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 22AB2
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Resveratrol; Piperine; Cerebral blood flow; Near- infrared spectroscopy; Bioavailability
MeSH Terms: interventions — Resveratrol; Silicon Dioxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 250mg trans- resveratrol (Experimental)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)
- 250mg trans-resveratrol with 20mg piperine (Experimental)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Trans- resveratrol; Other: Placebo (silica)

INTERVENTIONS:
Dietary Supplement: Trans- resveratrol — All 23 participants who completed the study took part in 3 conditions; receiving either 250mg resveratrol, 250mg resveratrol with 20mg piperine or placebo on separate days (with a 48hr-14 day wash-out period between each treatment) with the order dictated by Latin square. Treatment was in the form of powder and administered in capsule form, in a double blind manner.
Other: Placebo (silica) — All 23 participants who completed the study took part in 3 conditions; receiving either 250mg resveratrol, 250mg resveratrol with 20mg piperine or placebo on separate days (with a 48hr-14 day wash-out period between each treatment) with the order dictated by Latin square. Treatment was in the form of powder and administered in capsule form, in a double blind manner.

SUMMARY:
Resveratrol is associated with a plethora of physiological effects in humans, including modulation of cerebral blood flow, despite apparently poor bioavailability. This study investigated whether the physiological effects of resveratrol could be affected when co-supplemented with piperine, an alkaloid which may be able to enhance the bioavailability of resveratrol.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35 years old
* Healthy
* Non-smoker

Exclusion Criteria:

* Not proficient in English
* Taking medication or herbal supplements
* Pregnant or breast feeding
* Heavy caffeine consumer
* History of head trauma, migraines, learning difficulties, ADHD, gastrointestinal problems.
* Food allergies of intolerances

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Modulation of levels of total haemoglobin | 80 minutes following treatment administration
Modulation of levels of deoxygenated haemoglobin | 80 minutes following treatment administration
Modulation of levels of oxygenated haemoglobin | 80 minutes following treatment administration

SECONDARY OUTCOMES:
Number of participants displaying significant modulation of cognitive performance | 40-80 minutes post dose
  Cognitive performance was assessed at baseline and then again 40 minutes post-treatment to assess if any changes had taken place.

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Wightman, Principal Investigator — Northumbria University
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Wightman EL, Reay JL, Haskell CF, Williamson G, Dew TP, Kennedy DO. Effects of resveratrol alone or in combination with piperine on cerebral blood flow parameters and cognitive performance in human subjects: a randomised, double-blind, placebo-controlled, cross-over investigation. Br J Nutr. 2014 Jul 28;112(2):203-13. doi: 10.1017/S0007114514000737. Epub 2014 May 7. PMID 24804871